CLINICAL TRIAL: NCT01178528
Title: Effect of Ivabradine, Carvedilol or Their Combination in Patients With Heart Failure
Brief Title: Heart Rate Reduction in Heart Failure
Acronym: CARVIVA-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Giuseppe M.C. Rosano, Principal investigato, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTG001-07
Record Dates: First submitted 2010-04-19; First posted 2010-08-10 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Heart Failure
Keywords: heart failure; heart rate; ivabradine; carvedilol
MeSH Terms: conditions — Heart Failure | interventions — Ivabradine; Carvedilol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ivabradine (Experimental): 7.5 mg bd
  Interventions: Drug: ivabradine
- Carvedilol (Active Comparator): up to 25 mg bd
  Interventions: Drug: Carvedilol
- "Drug:Carvedilol" and "Drug:Ivabradine" (Experimental): up to 12.5/5 mg bd
  Interventions: Drug: "Drug:Carvedilol" and "Drug:Ivabradine"

INTERVENTIONS:
Drug: ivabradine — 7.5 mg bd
  Arms: Ivabradine
Drug: "Drug:Carvedilol" and "Drug:Ivabradine" — up to 12.5/5 mg bd
  Arms: "Drug:Carvedilol" and "Drug:Ivabradine"
Drug: Carvedilol — 25 mg bd
  Arms: Carvedilol

SUMMARY:
Patients with heart failure (HF) have a limited exercise tolerance,few pharmacological interventions have been proven effective in improving exercise capacity. At the presence there i conflicting evidence on the effectiveness of beta-blockers on exercise capacity. Ivabradine has been shown to improve prognosis in patients with ischemic heart disease, left ventricular dysfunction and heart rate > 70 bpm. The association of ivabradine and atenolol has been proven effective in increasing exercise tolerance in patients with ischemic heart disease. Aim of the present study is to evaluate the effect of heart rate reduction with ivabradine, carvedilol or their combination in patients with heart failure of ischemic origin.

DETAILED DESCRIPTION:
Patients with chronic heart failure of ischemic origin (120) Stable coronary artery disease Acute coronary syndromes > 3 months Revascularization procedures > 3 months Naive on heart rate reducing agents New York Heart Association (NYHA) Class II III 6 minute walking test (6MW) tolerance between 200 and 400 m Stable medications for the past 3 months

Treatment Ivabradine up to 7.5 mg b.i.d. Carvedilol up to 25 mg b.i.d. Carvedilol and Ivabradine up to 12.5/5 mg b.i.d.

Efficacy measure Intention to treat Exercise tolerance Quality of life

ELIGIBILITY:
Inclusion Criteria:

* heart failure II-III
* ischemic origin
* stable medications from at least 3 months
* > 3 months from an acute ischemic syndrome or revascularization procedure
* naive on heart rate reducing agents

Exclusion Criteria:

* bradycardia
* hypersensitivity or contraindications to study drugs
* exercise tolerance at 6 minute walking test <100 m or >400 m

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Volterrani, MD, Principal Investigator — IRCCS San Raffaele; Giuseppe MC Rosano, MD, PhD, Study Chair — IRCCS San Raffaele; Cristiana Vitale, MD, PhD, Study Director — IRCCS San Raffaele
Locations (2):
- Italy (2):
  - Centre for Clinical and Basic Research - IRCCS San Raffaele, Roma, Italy
  - IRCCS San Raffaele, Roma, Italy

REFERENCES:
- [Background] Fasullo S, Cannizzaro S, Maringhini G, Ganci F, Giambanco F, Vitale G, Pinto V, Migliore G, Torres D, Sarullo FM, Paterna S, Di Pasquale P. Comparison of ivabradine versus metoprolol in early phases of reperfused anterior myocardial infarction with impaired left ventricular function: preliminary findings. J Card Fail. 2009 Dec;15(10):856-63. doi: 10.1016/j.cardfail.2009.05.013. Epub 2009 Jul 3. PMID 19944362
- [Background] Swedberg K, Komajda M, Bohm M, Borer JS, Ford I, Tavazzi L. Rationale and design of a randomized, double-blind, placebo-controlled outcome trial of ivabradine in chronic heart failure: the Systolic Heart Failure Treatment with the I(f) Inhibitor Ivabradine Trial (SHIFT). Eur J Heart Fail. 2010 Jan;12(1):75-81. doi: 10.1093/eurjhf/hfp154. Epub 2009 Nov 5. PMID 19892778
- See also: European Society Cardiology guidelines — http://www.escardio.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Ivabradine: up to 7.5 mg b.i.d.
- Carvedilol: up to 25 mg b.i.d.
- Carvedilol and Ivabradine: up to 12.5 / 5 mg b.i.d.
Period: Overall Study
Arm/Group | Ivabradine | Carvedilol | Carvedilol and Ivabradine
Started | 41 | 38 | 42
Completed | 41 | 38 | 42
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivabradine | Carvedilol | Carvedilol and Ivabradine | Total
Number analyzed (Participants) | 41 | 38 | 42 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 32 | 91
  >=65 years | 11 | 9 | 10 | 30
Sex/Gender, Customized [Number; unit: participants]
  MALE | 28 | 26 | 28 | 82
  FEMALE | 13 | 12 | 14 | 39
Region of Enrollment [Number; unit: participants]
  Italy | 41 | 38 | 42 | 121
Exercise Tolerance Assessed by 6 Minute Walking Test [Mean (Standard Deviation); unit: meters] | 346.7 (112.0) | 379.0 (96.3) | 358.2 (107.6) | 361.3 (105.3)
Maximal Oxygen Consumption [Mean (Standard Deviation); unit: mL/Kg/min] | 12.05 (2.1) | 12.3 (2.6) | 12.4 (2.5) | 12.25 (2.4)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] | 4.3 (0.5) | 4.6 (0.8) | 4.7 (0.8) | 4.5 (0.7)
New York Heart Association (NYHA) class [Number; unit: participants] — The NYHA Classification system is a measure of functional status. Class II describes patients with cardiovascular disease (CVD) resulting in slight limitation of physical activity and comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain. There is objective evidence of minimal CVD. Class III describes patients with CVD resulting in marked limitation of physical activity and comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation, dyspnea, or anginal pain. There is objective evidence of moderately severe CVD.
  participants
    class II | 20 | 22 | 21 | 63
    class III | 21 | 16 | 21 | 58

OUTCOME MEASURES:

1. Primary Outcome: Exercise Tolerance Assessed by 6 Minute Walking Test
Description: Distance measured at 6 minute walking test. The 6 minute walking test was performed according to standardised procedure at baseline, before inclusion (at least 1 week after baseline evaluation), and at the end of the study. Patients who had not done at least two tests in the past underwent two practice 6 minute walking tests at least 3 days apart. Results are expressed in terms of distance walked (metres). The test was supervised by a physical therapist.
  Patients were asked to walk at their own maximal pace a 100 m long hospital corridor. At the beginning of the last (6th) minute of the test a standard phrase of encouragement was told. Patients were allowed to stop if signs or symptoms of significant distress occurred (dyspnea, angina), through they were instructed to resume walking as soon as possible.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ivabradine | Carvedilol | Carvedilol and Ivabradine
Number analyzed (Participants) | 41 | 38 | 42
meters | 474.8 (127.3) | 435.7 (121.3) | 453.1 (87.4)

2. Secondary Outcome: Quality of Life
Description: Quality of life (QoL) was evaluated using the Visual Analogue Scale (VAS) which is a global measurement of QoL, allowing a subjective assessment of the impact of the disease and treatment. Patients are asked to indicate their current state in a line from 0 (worst state) to 10 (best state), with higher values therefore representing a better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ivabradine | Carvedilol | Carvedilol and Ivabradine
Number analyzed (Participants) | 41 | 38 | 42
units on a scale | 6.7 (0.9) | 4.1 (0.6) | 6.1 (0.6)

3. Primary Outcome: Maximal Oxygen Consumption
Description: Functional capacity was assessed by means of a cardiopulmonary exercise test with a bicycle ergometer with gas exchange monitoring (Vmax 29 C, SensorMedics). Peak oxygen consumption was defined as the maximal oxygen consumption (MVO2) observed during exercise.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mL/Kg/min
Groups:
- Ivabradine: 7.5 mg b.i.d.
Arm/Group | Ivabradine | Carvedilol | Carvedilol and Ivabradine
Number analyzed (Participants) | 41 | 38 | 42
mL/Kg/min | 15.8 (1.9) | 12.9 (2.4) | 14.7 (1.6)

4. Secondary Outcome: New York Heart Association (NYHA) Class
Description: The 1994 NYHA Classification system is a measure of functional status. It was designed for clinical assessment of patients by physicians as NYHA class I, II, III, or IV, on the basis of patient's limitations in physical activities caused by cardiac symptoms.
  Class I describes patients with cardiovascular disease (CVD) but without resulting limitation of physical activity. There is no objective evidence of CVD.
  Class II describes patients with CVD resulting in slight limitation of physical activity. There is objective evidence of minimal CVD.
  Class III describes patients with CVD resulting in marked limitation of physical activity. There is objective evidence of moderately severe CVD.
  Class IV describes patients with CVD resulting in inability to carry on any physical activity without discomfort. There is objective evidence of severe CVD.
  Here we report data on number of patients showing an improvement by at least one NYHA class according to treatment allocation.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Ivabradine | Carvedilol | Carvedilol and Ivabradine
Number analyzed (Participants) | 41 | 38 | 42
participants | 30 | 5 | 20

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Ivabradine | Carvedilol | Carvedilol and Ivabradine
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/38 | 0/42
Other Adverse Events (participants affected / at risk) | 0/41 | 0/38 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes